CLINICAL TRIAL: NCT04811118
Title: A Randomized, Open-label, Two-period, Crossover Trial to Compare the Pharmacokinetic Profiles Between Albumin-bound Docetaxel and Taxotere in Patients With Advanced Solid Tumors
Brief Title: The Comparison of the Pharmacokinetics of Albumin-bound Docetaxel and Taxotere
Status: Unknown | Phase: Phase 1 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: CSPC ZhongQi Pharmaceutical Technology Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Treatment
Other Study IDs: HB1801-CSP-002
Record Dates: First submitted 2021-03-10; First posted 2021-03-23 (Actual); Last update posted 2022-01-31 (Actual); Status verified 2021-06

CONDITIONS: Advanced Solid Tumors
MeSH Terms: interventions — Docetaxel; Injections

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Albumin-bound docetaxel (Experimental): Subjects will receive albumin-bound docetaxel via intravenous infusion (IV) once every three weeks (a cycle), at the dose of 75mg/m2
  Interventions: Drug: Docetaxel for Injection (Albumin-bound)
- Taxotere (Experimental): Subjects will receive Taxotere via intravenous infusion once every three weeks (a cycle), at the dose of 75mg/m2.
  Interventions: Drug: Taxotere

INTERVENTIONS:
Drug: Docetaxel for Injection (Albumin-bound) — Docetaxel for Injection (Albumin-bound) by intravenous infusion
  Other Names: Docetaxel
  Arms: Albumin-bound docetaxel
Drug: Taxotere — Taxotere
  Other Names: Docetaxel
  Arms: Taxotere

SUMMARY:
This is a randomized, open-label, two-period, crossover trial to evaluate the pharmacokinetic profiles of albumin-bound docetaxel for intravenous infusion and Taxotere in patients with advanced solid tumors.

DETAILED DESCRIPTION:
The trial will be performed as a randomized, open-label, two-period crossover trial to compare the test drug (T, albumin-bound docetaxel) to the reference drug (R, Taxotere). Approximately 28 subjects will be randomized to the two treatment sequences (T-R or R-T) at the ratio of 1:1. Each enrolled subject will receive an intravenous infusion of the reference drug and the test drug in two treatment periods per the randomization schedule. The treatment periods will be separated by a washout period of 21 to 35 days. After completing two cycles of treatments, subjects may continue to receive the treatment used in the second cycle according to the responses (up to 1 year).

ELIGIBILITY:
Inclusion Criteria:

1. Age ≥18, ≤65 years, no gender limitation；
2. Histologically or cytologically confirmed diagnosis of advanced or metastatic solid tumors, for which standard therapy either does not exist or has proven to be ineffective, intolerable, unacceptable or with other limitations for the patient；
3. At least one measurable lesion as per RECIST version 1.1；
4. Eastern Cooperative Oncology Group (ECOG) Performance Status (PS) 0 or 1；
5. Life expectancy ≥3 months；
6. Major organ function within 7 days prior to treatment meets the following criteria (no blood transfusion, EPO, G-CSF or other medical support within 14 days prior to study drug administration): ANC≥1.5×109/L，PLT≥100×109/L，Hb≥90g/L or≥5.6 mmol/L；Cr≤1.5×ULN and creatinine clearance rate≥50ml/min；TBIL≤1.0×ULN，AAG≥1.0×LLN，except for those with AST/ALT>1.5 × ULN and ALP>2.5× ULN;
7. Patients of childbearing potential must agree to use effective contraceptive measures (such as IUD, contraceptive pill or condom) during the period of the trial and for at least 6 months after completion of the study. Female patients must be negative on the serum pregnancy test within 7 days before enrollment, and must be nonlactating. Male patients refrains from donating sperm during the study period and for at least 6 months after completion of the study；
8. Signed informed consent form.

Exclusion Criteria:

1. Treatment failure of prior docetaxel or paclitaxel treatment (such as: patients who relapse within 6 months after last treatment);
2. Chemotherapy, radiotherapy, biotherapy, endocrine therapy, targeted therapy, immunotherapy and other anti-tumor treatment within 4 weeks of the first dose of the study drug, 6 weeks for mitomycin C or nitrosoureas, 2 weeks (or 5 half-lives whichever is longer) for using fluorouracil or small molecule targeted drugs, 2 weeks for using traditional Chinese medicine with anti-tumor indications；
3. Currently enrolled in any other clinical study, or administration of other investigational agents within 4 weeks of the first dose of the study drug；
4. Major surgery (excluding biopsy) or significant trauma within 4 weeks of the first dose of the study drug. Or have a surgical schedule during the study period.
5. Administration of glucocorticoids or other immunosuppressants within 14 days prior to the first dose of d the study drug.Local, ocular, intraarticular, intranasal, inhaled glucocorticoids, and a short-term use of glucocorticoids for preventive treatment is allowed；
6. Concomitant use of strong CYP3A4 inhibitors or inducers within 14 days of the first dose of the study drug；
7. Allergic history to Taxanes or any excipients of the study drug (CTCAE 5.0 grade ≥ 3 grade)；
8. Adverse reactions from the previous anti-tumor treatment have not yet recovered to ≤ level 1 based on CTCAE 5.0 (except for the toxicity without safety risk judged by the investigator, such as hair loss)；
9. Central nervous system metastasis or meningeal metastasis with clinical symptoms, or other evidence shows that the patient's central nervous system metastasis or meningeal metastasis has not been controlled and not suitable for the study according to the judgment of the investigator；
10. History of autoimmune diseases, immunodeficiency, including HIV positive, or other acquired, congenital immunodeficiency, or organ transplant history；
11. Known Hepatitis B Virus (HBV), Hepatitis C Virus (HCV), or other active viral infection；
12. History of serious cardiovascular disease；
13. Uncontrollable effusion (eg. large amount of pleural effusion, ascites or pericardial effusion)；
14. Known alcohol or drug abuse；
15. Visual impairment such as cystoid macular edema；
16. History of neurological or psychiatric disorders；
17. Homozygous carriers of ABCB1-1236C>T（rs1128503）;
18. Not suitable for this study as determined by the investigator due to other reasons.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 27 (Actual)
Dates: Start 2021-05-18 (Actual); Primary Completion 2022-10-31 (Estimated); Study Completion 2022-12-31 (Estimated)

PRIMARY OUTCOMES:
The pharmacokinetic parameters (free docetaxel and total docetaxel) : Cmax | At the end of Cycle 2 (each cycle is 21 days)
  Peak Plasma Concentration (Cmax)
The pharmacokinetic parameters (free docetaxel and total docetaxel) : AUC0-t、AUC0-∞ | At the end of Cycle 2 (each cycle is 21 days)
  Area under the plasma concentration versus time curve (AUC)

SECONDARY OUTCOMES:
1.The occurrence and frequency of adverse events and serious adverse events | through study completion, up to 18 weeks
  1. The occurrence and frequency of adverse events and serious adverse events
2. 1 Efficacy measures such as overall response rate (ORR) | through study completion, up to 18 weeks
  overall response rate (ORR)
2. 2 Efficacy measures such as progression-free survival (PFS) | through study completion, up to 18 weeks
  progression-free survival (PFS)
2.3 Efficacy measures such as disease control rate (DCR) | through study completion, up to 18 weeks
  disease control rate (DCR)
2. 4 Efficacy measures such as duration of response (DOR). | through study completion, up to 18 weeks
  duration of response (DOR)

CONTACTS AND LOCATIONS:
Overall Officials: Hui Shan, master, Study Director — CSPC ZhongQi Pharmaceutical Technology Co., Ltd.
Locations (1):
- Cangzhou Central Hospital, Cangzhou, China